CLINICAL TRIAL: NCT06227962
Title: Cognitive Functioning and Health Related Quality of Life in Retinoblastoma Survivors (8-35 Years): The Role of Cancer Treatment and Repeated Anesthesia
Brief Title: Cognitive Functioning and Health Related Quality of Life in Retinoblastoma Survivors
Acronym: RbNeuroQoL
Status: Enrolling by invitation | Type: Observational
Sponsor: Amsterdam University Medical Center (Other)
Responsible Party: Principal Investigator, Annette Moll, M.D., PhD, Clinical professor, Amsterdam University Medical Center
Organization: Amsterdam UMC, location VUmc (Other)
Other Study IDs: NL82126.029.22; SKOCA 2009020 (Other Grant/Funding Number: Stichting Kinderoncologisch Centrum Amsterdam); Uitzicht 2021-13-Moll (Other Grant/Funding Number: UitZicht (a cooperation of several Dutch funds))
Record Dates: First submitted 2023-12-20; First posted 2024-01-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Retinoblastoma; Neurocognitive Dysfunction; Health-Related Behavior
Keywords: Retinoblastoma; Cognition; Psychosocial functioning; HRQoL
MeSH Terms: conditions — Retinoblastoma; Cognition Disorders; Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retinoblastoma Survivors: Children and adults who survived retinoblastoma (8-35 years of age)
  Interventions: Diagnostic Test: Neuropsychological assesment; Diagnostic Test: Psychosocial functioning and quality of life (questionnaires)
- Retinoblastoma Risk Carriers: Children and adults who (might) carry a genetic risk to develop retinoblastoma (8-35 years of age)
  Interventions: Diagnostic Test: Neuropsychological assesment; Diagnostic Test: Psychosocial functioning and quality of life (questionnaires)
- Parents: Parents of Rb patients, Rb survivors, or Rb risk carriers (6 months-12 years of age)
  Interventions: Diagnostic Test: Parental psychosocial functioning (questionnaires)

INTERVENTIONS:
Diagnostic Test: Neuropsychological assesment — Estimated intelligence (subtasks of Wechsler Intelligence Scale for Children - Fifth edition -Dutch version [WISC-V-NL] or Wechsler Adult Intelligence Scale - Forth edition - Dutch version [WAIS-IV-NL]); Vienna reaction time; Rey auditory verbal learning test; Word fluency; Beery-Buktenica Developmental Test of Visual-Motor Integration, 6th Edition; Test of Everyday Attention for Children (TEA-Ch), subtask Score!/ or Test of Everyday Attention (TEA), subtask Elevator task; Trail making test; Word-color interference test
  Groups: Retinoblastoma Risk Carriers; Retinoblastoma Survivors
Diagnostic Test: Psychosocial functioning and quality of life (questionnaires) — Anxiety (PROMIS); Depression (PROMIS); Peer-interaction (PROMIS); Perceived neurocognitive functioning (PROMIS); Participation and activity (PAY-CY); Trauma (KJTS/PCL-5); Health related quality of life (PEDSQL)
  Groups: Retinoblastoma Risk Carriers; Retinoblastoma Survivors
Diagnostic Test: Parental psychosocial functioning (questionnaires) — Anxiety (PROMIS); Depression (PROMIS); Distress Thermometer-Parents (DT-P); Trauma (PCL-5)
  Groups: Parents

SUMMARY:
A retrospective crosssectional observational study of the effects of oncological treatment and frequent general anesthesia on neuropsychological development, psychosocial functioning (in terms of anxiety, depression, peer relations, perceived cognitive functioning and potential trauma) and health related quality of life in children and young adults who were treated or screened for retinoblastoma.

DETAILED DESCRIPTION:
Retinoblastoma (Rb) is the most common form of ocular cancer in children, with high survival rates in developed countries (>90%). Rb can develop unilateral (one eye affected, sometimes hereditary), or bilateral (both eyes, always hereditary). Children are usually diagnosed at a young age (<5 years) and are subjected to an intensive treatment and follow-up protocol immediately after. If Rb is diagnosed in early disease stages, eye-saving treatment could be provided, such as laser, cryo-, chemotherapy and/or radiotherapy -or a combination of these. When discovered in a later disease stage, enucleation (removing the eye) is often inevitable. Brothers and sisters or offspring of heredity Rb survivors that are at risk to develop Rb themselves (so called 'Rb risk carriers') will be screened according to the Dutch Rb Screening Protocol. The medical treatment and follow-up of Rb patients and screening of Rb risk carriers takes place under general anesthesia (GA) up to four or five years of age. At this age the brain is still developing and therefore extra vulnerable to iatrogenic damage, including neuropsychological complications. Immediate effects of the oncological treatment, as well as secondary effects due to multiple GA on cognitive development in Rb survivors is still understudied. Rb survivors report disease-related limitations in daily life and lower health related quality of life (HRQoL), which might be related to impaired cognitive functioning. Apart from possible immediate or secondary treatment effects, children with Rb are known to be experiencing psychosocial struggles, including anxiety and depression, declined participation and/or pediatric trauma, which may negatively affect HRQoL as well. Despite the impact on general wellbeing and HRQoL, the cognitive and emotional aspects of Rb are largely under addressed in pediatric care. It is important to gain insight in the cognitive development and psychosocial functioning from childhood into young adulthood of Rb survivors, as well psychosocial functioning of the parents in order to provide timely interventions, minimizing possible long-term consequences. It is hypothesized that extensive treatment and multiple GA is negatively associated with cognitive functioning, psychosocial functioning and HRQoL in Rb survivors and Rb risk carriers. Moreover, that psychological struggles and/or trauma strengthen these associations.

ELIGIBILITY:
Inclusion Criteria Rb survivors and Rb risk carriers (age 8-35 years):

* Rb diagnosis, (main) treatment and follow-up of Rb patients and -survivors, or Rb screening took place at the Dutch Retinoblastoma Expertise Center of the Amsterdam University Medical Center,
* Rb survivor or former Rb risk carriers is between 8 and 35 years old,
* Average understanding of the Dutch language.

Inclusion Criteria parents of Rb patients, Rb survivors or Rb risk carriers (6 months - 12 years):

* Being a caregiver of a Rb survivor or Rb risk carrier that have been diagnosed and receive(d) (main) treatment and follow-up or screening at the Dutch Retinoblastoma Expertise Center of the Amsterdam University Medical Center,
* The related Rb survivor or Rb risk carrier is < 12 years old,
* Average understanding of the Dutch language.

Exclusion Criteria:

* Pre-existing documented developmental delay and/or severe cognitive impairments (IQ <70),
* Having an active, uncontrolled psychiatric illness,
* Rb diagnostic trajectory, treatment and follow-up at another hospital or before the founding of the Dutch Retinoblastoma Expertise Center in 1991. With exception of Rb survivors (diagnosed >1991) who apart from treatment at the Dutch Retinoblastoma Center also required specialized treatment (such as radiation) at another center: they are illegible for inclusion.

Ages: 6 Months to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Approximately 350 Rb survivors and 310 Rb risk carriers (<35 years) that have been treated or screened at the Dutch Retinoblastoma Expertise Center of the Amsterdam University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Estimated intellectual functioning (Neurocognition) | This concerns a cross-sectional study meaning that a neuropsychological assessment is carried out only once on all participants during the course of the study until study completion, approximately in 2027.
  Is assessed using 2 or 4 subtasks of the Dutch translation of the Wechsler Intelligence Scale for Children-Fifth edition (WISC-V-NL [8-16 years]) or the Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV-NL [16-35 years]), depending on the visual ability of the participant.
  The 'Verbal Comprehension Index' (VCI) is assessed in all participants using the verbal subtests 'Similarities' and 'Vocabulary'. The 'Perceptual Reasoning Index' (PRI) is assessed in all sighted participants using the subtests 'Matrix Reasoning' and 'Block Design'.
  Index scores are calculated (range 55-145; M=100, SD=10) and outcomes between 90-110 are considered average, <89 below average to borderline and >110 above average to highly gifted. Subscale outcomes (range 0-20; M=10, SD=2) between 8-12 are considered average, <8 below average, and >12 above average.
Processing speed (Neurocognition) | This concerns a cross-sectional study and data will be collected until April 2027. The neuropsychological assessment is carried out only once on all participants during the course of the study until study completion.
  Vienna S2 'Auditory Reaction Time' is only assessed in all participants. Additionally, Vienna S1 'Visual Reaction Time' and S3 'Combined [visual-auditory] Reaction Time', and subtasks 'Digital Symbol Coding' and 'Symbol Search' of the WISC-V-NL or WAIS-IV-NL will be assessed in sighted participants as well. Outcomes of the VTS will be calculated in T-Scores (range 20-80; M=50, SD=10), where a T-score between 40 and 60 is considered average, <40 below average and >60 above average. A WISC-V-NL or WAIS-IV-NL Index score will be calculated (range 55-145; M=100, SD=10) and is considered average between 90-110, <89 as below average to borderline, and >110 as above average to highly gifted. Subscale outcomes (range 0-20) between 8-12 are considered average, <8 below average and >12 above average.
Memory (Neurocognition) | This concerns a cross-sectional study and data will be collected until April 2027. The neuropsychological assessment is carried out only once on all participants during the course of the study until study completion.
  In all participants, encoding and retrieval of verbal information will be assessed using the Rey- Auditory Verbal Learning Test (RAVLT). Working memory will be assessed using the subtests 'Digit Span' of the WISC-V-NL (8-16 years) or WAIS-IV-NL (17-35 years) resulting in the 'Working Memory Index' (WMI).
  RAVLT outcomes will be calculated in T-Scores (range 20-80), where a T-score between 40 and 60 is considered average, <40 below average and >60 above average. WISC-V-NL or WAIS-IV-NL Index scores will be calculated (range 55-145; M=100, SD=10) and outcomes between 90-110 are considered average, <89 below average to borderline and >110 above average to highly gifted. Subscale outcomes (range 0-20; M=10, SD=2) between 8-12 are considered average, <8 below average, and >12 above average.
Verbal fluency (Neurocognition) | This concerns a cross-sectional study and data will be collected until April 2027. The neuropsychological assessment is carried out only once on all participants during the course of the study until study completion.
  Verbal fluency will be assessed in all participants using the Semantic condition of the Dutch translation of the subtask Word Production of the Developmental Neuropsychological Assessment (NEPSY-III-NL [age 8-12 years]) or the Word Fluency Test (WFT [13-35 years]), a Dutch translation of the Controlled Oral Word Association Test (COWAT)).
  NEPSY-III-NL outcomes will be calculated in norm scores (range 0-20; M=10, SD=2), where outcomes between 8-12 are considered average, <8 below average and >12 above average. Outcomes of the WFT will be calculated in T-Scores (range 20-80; M=50, SD=10), were a T-score between 40 and 60 is considered average, <40 below average, and >60 above average.
Visual Motor Integration (Neurocognition) | This concerns a cross-sectional study and data will be collected until April 2027. The neuropsychological assessment is carried out only once on all participants during the course of the study until study completion.
  Visual Motor Integration will be assessed in sighted participants only, using the Visual-Motor Integration (VMI), Visual Perception (VP) and Motor Coordination (MC) of the Beery-Buktenica Developmental Test of Visual-Motor Integration, 6th Edition, Beery-VMI.
  Standard scores (range 48-155; Mean=100, SD=15) will be calculated, as well as T-scores (range 55-145; M=50, SD=10). Standard scores between 85-115 are considered average, <85 below average to borderline, and >115 above average to highly gifted. T-scores between 40 and 60 are considered average, <40 below average, and >60 above average.
Sustained Auditory Attention (Neurocognition) | This concerns a cross-sectional study and data will be collected until April 2027. The neuropsychological assessment is carried out only once on all participants during the course of the study until study completion.
  Sustained auditory attention will be assessed in all participants using the subtask Score! of the Test of Everyday Attention for Children (TEA-Ch [6-16 years]; Publication date 2004) or the Elevator task of the Test of Everyday Attention (TEA [17-35 years]; Publication date 1994). Regarding the TEA-Ch, norm scores (range 1-19; M=10, SD=2) will be calculated, whereas outcomes between 8-12 are considered average, <8 below average, and >12 above average. The Elevator task of the TEA has 7 subsets, the participants receives one point per correct subset (max=7). An outcome of 7 is considered 'Normal', 6 is considered 'Subclinical Abnormal', and <5 is considered 'Clinical Abnormal'.
Executive functioning (Neurocognition) | This concerns a cross-sectional study and data will be collected until April 2027. The neuropsychological assessment is carried out only once on all participants during the course of the study until study completion
  The Executive functioning (EF) tasks will be assessed in sighted participants only. The Stroop Color Word Test of the Delis-Kaplan Executive Function System (D-KEFS; Publication date 2007) measures selective visual attention, cognitive flexibility, inhibition and processing speed. The Trail Making Test (TMT) of the D-KEFS (publication data 2007) assesses attention, visual screening and cognitive flexibility. Scale scores will be calculated (range 0-20; M-10, SD=2) and scores between 8-12 are considered average, scores <8 are considered below average, and scores >12 above average.
Anxiety (Psychosocial functioning) | This concerns a cross-sectional study. Digital questionnaires will be assessed (if applicable) within two weeks of the neuropsychological assessment, only once on all participants during the course of the study until study completion (expected 2027).
  Anxiety (proxy 5-16 years and self-report 8-35 years) is assessed using a digital Patient Reported Outcomes Measurement Information System (PROMIS), computer adaptive testing (CAT) questionnaire (using the Dutch KLIK portal [in Dutch Kwaliteit van Leven in Kaart/Mapping Quality of Life]). A standard Total Scale score (range 0-100) of 0-59 indicate no anxiety symptoms, between 60-69 subclinical anxiety symptoms, and >70 clinical anxiety symptoms.
Depression | This concerns a cross-sectional study. Digital questionnaires will be assessed (if applicable) within two weeks of the neuropsychological assessment, only once on all participants during the course of the study until study completion (expected 2027).
  Depression (proxy 5-16 years and self-report 8-35 years) is assessed using a digital PROMIS-CAT questionnaire (using the Dutch KLIK portal). A Standard Total Scale score (range 0-100) of 0-59 indicate no depression symptoms, between 60-69 subclinical depression symptoms, and >70 clinical depression symptoms.
Peer interaction (Psychosocial functioning)) | This concerns a cross-sectional study. Digital questionnaires will be assessed (if applicable) within two weeks of the neuropsychological assessment, only once on all participants during the course of the study until study completion (expected 2027).
  Peer interaction (self-report 9-17 years) is assessed using a digital PROMIS-CAT questionnaire (using the Dutch KLIK portal). A Standard Scale score (range 0-100) is calculated and outcomes. A norm score of <29 is considered having poor peer relations, between 29 and 39 suboptimal peer relations, and >39 having no peer relation problems.
Perceived neurocognitive functioning (Psychosocial functioning) | This concerns a cross-sectional study. Digital questionnaires will be assessed (if applicable) within two weeks of the neuropsychological assessment, only once on all participants during the course of the study until study completion (expected 2027).
  Perceived neuropsychological functioning (self-report 8-35 years) is assessed using a digital PROMIS-CAT questionnaire (using the Dutch KLIK portal). The questionnaire consists of 7 questions related to perceived problems regarding attention, focus, memory and reading comprehension. Questions are answered on a 4-point Likert scale (1=never, 2=sometimes, 3=often, 4=most of the time).
  Due to absence of standard data, standardized outcomes cannot be calculated. Outcomes of participants will be compared to each other, with a low score indicating good perceived cognitive functioning and a high score indicating declined perceived cognitive functioning
Participation and Activity (Psychosocial functioning) | This concerns a cross-sectional study. Digital questionnaires will be assessed (if applicable) within two weeks of the neuropsychological assessment, only once on all participants during the course of the study until study completion (expected 2027).
  Participation and activity (proxy 0-16 years and self-report 8-35 years) is assessed using the digital questionnaire Participation and Activity Inventory for Children and Youth (PAY-CY, publication date 2019, [using the Dutch KLIK portal]). Due to absence of standard data, outcomes (range 0-100) of participants will be compared to each other, with a high score indicating the absence of or fewer obstacles to activity and participation in daily life and a low score indicates much perceived obstacles. Outcomes relate to 'Activity and participation'. Additionally, 'Sensory functioning' and 'Parental component' is also assessed in the proxy questionnaires.
Trauma (psychosocial functioning) | This concerns a cross-sectional study. Digital questionnaires will be assessed (if applicable) within two weeks of the neuropsychological assessment, only once on all participants during the course of the study until study completion (expected 2027).
  Post-traumatic stress disorder (PTSD; proxy 3-16 years/ self-report 8-35 years) is assessed using the Dutch translation of the Child and Adolescent Trauma Screener (KJTS, in Dutch: Kind en Jeugd Trauma Screener [3-18 years]) or the PTSD Checklist for the DSM-5 (PCL-5 [18-35 years] using the Dutch KLIK portal)).
  Standard outcomes of the KJTS (range 0-60) regards 'Total Score', whereas <15 is considered within normal limits, 15-19 subclinical development of PTSD and >20 clinical development of PTSD. Regarding PCL-5, participants report a traumatic event ('Criteria A'). Standard outcomes are calculated in a 'Total Score' and sub scores corresponding to the DSM-5 criteria: 'Criteria B' (intrusive symptoms), 'Criteria C' (persistent avoidance), 'Criteria D' (negative alterations), and 'Criteria E' (arousal and reactivity). A Total Score (range 0-80) between 0-27 indicates no PTSD symptoms, between 28-32 subclinical PTSD development, and a total score of >33 development of clinical PTSD.
Health related quality of life (Psychosocial functioning) | This concerns a cross-sectional study. Digital questionnaires will be assessed (if applicable) within two weeks of the neuropsychological assessment, only once on all participants during the course of the study until study completion (expected 2027).
  Health Related Quality of Life (HRQoL; proxy 0-16 years and self-report 8-35 years) is assessed using the digital questionnaires Preschool Children's Quality of Life questionnaire (TAPQOL [0-2 years]) or Pediatric Quality of Life Inventory (PedsQL [3-35 years] using the Dutch KLIK portal)). All outcomes (range 0-100) will be compared to Dutch norm reference data (bases on age and gender) and cut off scores differ among age. High scores indicate good functioning. A deviation of 10 points below the national average score of same-sex peers is clinically relevant. Subscales of the TAPQOL relates to 'Stomachache', 'Skin Problems', 'Respiratory Problems', 'Sleeping Problems', 'Apatite', 'Positive mood', 'Anxiety', 'Livelihood' and 'Problem behavior'. Subscales of the PedsQL relate to the domains 'Physical Functioning' , 'Emotional Functioning', 'Social Functioning' and 'School functioning'.
Study specific outcomes | This concerns a cross-sectional study. Digital questionnaires will be assessed (if applicable) within two weeks of the neuropsychological assessment, only once on all participants during the course of the study until study completion (expected 2027).
  Four questions were asked to all participants:
  1. Satisfaction with physical appearance, measured on a scale of 0-10 where 0 indicates completely dissatisfied and 10 indicates very satisfied.
  2. Whether the participant has been under anesthesia for conditions other than retinoblastoma and if so, how often. (open end)
  3. Whether the participant has been diagnosed with a psychiatric (DSM-5) disorder. (open end)
  4. An open end question whether the participant would like to add or mention anything the participant considers worth mentioning.

SECONDARY OUTCOMES:
Parental anxiety | This concerns a cross-sectional study. The digital questionnaires will be assessed only once on all parents of participants (age 0-12) during the course of the study until study completion, expected in 2027.
  Parental anxiety is assessed using a digital PROMIS-CAT questionnaire (using the Dutch KLIK portal). Standard outcomes (range 0-100) between 0-59 indicate no anxiety symptoms, between 60-69 subclinical anxiety symptoms, and >70 clinical anxiety symptoms.
Parental depression | This concerns a cross-sectional study. The digital questionnaires will be assessed only once on all parents of participants (age 0-12) during the course of the study until study completion, expected in 2027.
  Parental depression is assessed using a digital PROMIS-CAT questionnaire (using the Dutch KLIK portal). Standard outcomes (range 0-100) between 0-59 indicate no depression symptoms, between 60-69 subclinical depression symptoms, and >70 clinical depression symptoms.
Parental symptoms of distress | This concerns a cross-sectional study. The digital questionnaires will be assessed only once on all parents of participants (age 0-12) during the course of the study until study completion, expected in 2027.
  Is assessed using the digital Distress Thermometer for Parents (DT-P) questionnaire (using the Dutch KLIK portal). Total perceived stress is rated on a 10 points scale (0=no distress, 10=maximum distress). Domain scores will be calculated, which relate to: 'Practical Functioning', 'Social Functioning', 'Emotional Functioning', 'Physical Functioning', 'Cognitive Functioning', and 'Child-parent Interaction and Upbringing'. High scores on the subdomains indicate higher levels of distress, low scores indicate low levels of distress. Additionally, four questions addresses amount of perceived support, perceived recognition by others, whether the parent is chronically ill itself, and about experience with the medical staff. whether they received supported care by family or professional help and the need to consult a healthcare professional.
Parental trauma | This concerns a cross-sectional study. The digital questionnaires will be assessed only once on all parents of participants (age 0-12) during the course of the study until study completion, expected in 2027.
  Parental trauma related to retinoblastoma (diagnosis, treatment and/or follow-up) is assessed using the Dutch translation of the digital questionnaire PTSD Checklist for the DSM-5 (PCL-5). Parents complete 20 questions related to their child's illness (i.e. (risk of) retinoblastoma) ('Criteria A'). Standard outcomes are calculated in a 'Total Score' and sub scores corresponding to the DSM-5 criteria: 'Criteria B' (intrusive symptoms), 'Criteria C' (persistent avoidance), 'Criteria D' (negative alterations), and 'Criteria E' (arousal and reactivity). A Total Score (range 0-80) between 0-27 indicates no PTSD symptoms, between 28-32 indicates subclinical PTSD development, and a total score of >33 indicates development of clinical PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Annette C. Moll, MD PhD, Principal Investigator — Amsterdam University Medical Center
Locations (1):
- Amsterdam University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Datasets and statistical codes of the study will be made available upon request to the international science and rehabilitation community